CLINICAL TRIAL: NCT06375122
Title: Natural History Study of Kaposi Sarcoma
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001951; 001951-C
Record Dates: First submitted 2024-04-18; First posted 2024-04-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-04-22

CONDITIONS: Kaposi Sarcoma; HIV
Keywords: Kaposi Sarcoma; Samples and data collection; Longitudinal clinical evaluations
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with Kaposi sarcoma

SUMMARY:
Background:

Kaposi sarcoma (KS) is a type of tumor caused by the Kaposi sarcoma herpesvirus. KS usually affects the skin, but lesions can also appear in the lymph nodes, lungs and digestive tract. KS is most common in people with compromised immunity, but it also appears in otherwise healthy people. Researchers want to understand more about how KS develops, why it may recur, and how it affects the immune system and organs.

Objective:

To learn more about the natural history of KS.

Eligibility:

People aged 18 years and older with KS.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have an imaging scan. They may need a new biopsy: Tissue samples may be cut from their tumor. Their ability to perform normal activities will be assessed.

Participants will visit the clinic to have their KS evaluated. In addition to the imaging scans and other tests performed during screening, procedures may include:

Eye exam.

Ultrasound exam of the heart (electrocardiogram).

Collection of saliva and urine samples.

Biopsies of the skin or lymph nodes.

Swabs of the anus and cervix.

Photographs of skin lesions.

Removal of fluid samples from the space around the lungs, intestine, or heart.

The evaluation visit will be repeated 5 more times over 18 months and then yearly for up to 10 years.

Participants will follow their standard treatment for KS during the study.

DETAILED DESCRIPTION:
Background:

* Kaposi sarcoma (KS) is a multicentric angioproliferative tumor caused by Kaposi sarcoma herpesvirus (KSHV) that most frequently involves skin, but can also involve lymph nodes, lungs, and gastrointestinal tract. It is most common in people with human immunodeficiency virus (HIV) or other forms of immune compromise.
* Patients with HIV-associated KS have worse survival than HIV-infected patients without KS.
* KS can occur alone or with other KSHV-associated disorders such as multicentric Castleman disease (MCD), primary effusion lymphoma (PEL), or KSHV-associated inflammatory cytokine syndrome (KICS).
* The natural history of KS is incompletely understood as it occurs in different epidemiologic subtypes (including those with HIV, particularly among individuals with well-controlled HIV and robust CD4 T cell counts, and those who are HIV-negative).
* The longitudinal evaluations along with tissue sample collection, imaging studies, and participant reported outcomes will allow for the development of a better understanding of the natural history of this disease, and the development of the basis for more effective treatments.

Objective:

-To characterize the natural history of KS, including presentation, manifestation, and proportion of participants with KS with remission and recurrence by epidemiologic subtype

Eligibility:

* Participants with histologically confirmed KS
* Age >=18 years
* No active KICS or MCD

Design:

* This will be a long-term trial to comprehensively study participants with KS.
* Medical history including HIV characteristics, research specimens such as KS tissue, blood and saliva will be obtained through the course of KS management with specific attention to patterns related to disease recurrence and progression, response to therapies, and duration of response.
* Outcomes and factors that influence the onset and persistence of KS over the natural history of this condition will be explored in collaboration with other centers that treat participants with KS.
* We anticipate accruing 230 participants on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must have histological KS confirmed by the Laboratory of Pathology (LP), NCI.

* KS as assessed by cutaneous or oral KS lesions or other assessable KS disease.
* Age >=18 years.
* ECOG performance status <=4.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants with active KSHV-associated inflammatory cytokine syndrome (KICS), multicentric Castleman disease (MCD), or primary effusion lymphoma (PEL).
* Participants with serious and/or uncontrolled severe intercurrent illness, such as opportunistic infections, that in the judgement of the investigator would preclude participation in the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Kaposi sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize the natural history of Kaposi sarcoma (KS), including presentation, manifestation, and proportion of participants with KS with remission and recurrence by epidemiologic subtype | 10 years
  Assessment of the proportion of participants with KS by epidemiologic subtype who experience remission and recurrent KS over the course of the disease

SECONDARY OUTCOMES:
To evaluate differences in rates of KS recurrence by human immunodeficiency virus (HIV) status and CD4 T cell count | 10 years
  Assess the proportion of recurrence by HIV status and by CD4 T cell count.
To evaluate the emergence of KSHV-associated inflammatory syndromes in the natural history of KS | 10 years
  Evaluate the proportion of participants with the emergence of KICS, MCD and/or PEL during the course of the natural history evaluation. Evaluation of parameters of CBC, acute, hepatic, mineral panels and CRP may provide predictive markers for the emergence of these conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Bhutani M, Polizzotto MN, Uldrick TS, Yarchoan R. Kaposi sarcoma-associated herpesvirus-associated malignancies: epidemiology, pathogenesis, and advances in treatment. Semin Oncol. 2015 Apr;42(2):223-46. doi: 10.1053/j.seminoncol.2014.12.027. Epub 2014 Dec 31. PMID 25843728
- [Background] Robbins HA, Pfeiffer RM, Shiels MS, Li J, Hall HI, Engels EA. Excess cancers among HIV-infected people in the United States. J Natl Cancer Inst. 2015 Feb 6;107(4):dju503. doi: 10.1093/jnci/dju503. Print 2015 Apr. PMID 25663691
- [Background] Ballon G, Akar G, Cesarman E. Systemic expression of Kaposi sarcoma herpesvirus (KSHV) Vflip in endothelial cells leads to a profound proinflammatory phenotype and myeloid lineage remodeling in vivo. PLoS Pathog. 2015 Jan 21;11(1):e1004581. doi: 10.1371/journal.ppat.1004581. eCollection 2015 Jan. PMID 25607954
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001951-C.html